CLINICAL TRIAL: NCT05946070
Title: Effectiveness of Mobile Based Monitoring System in the Management of Chemotherapy-Related Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gulbeyaz Can, Professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 35621
Record Dates: First submitted 2023-06-22; First posted 2023-07-14 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Cancer; Chemotherapeutic Toxicity; Mobile Applications
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (ONKOSIS) (Experimental): Patients in the intervention group will be instructed to use the mobile application. Patients in the experimental group will be able to access the application contents without restrictions and will be able to use the in-app messaging module as well as the risk factors, symptom findings, and intervention suggestions for symptom management.
  Interventions: Other: ONKOSIS
- Control group (No Intervention): Patients in the control group will receive standard care as is currently available at their clinical site. They will use demo version of the mobile application only for assessing symptom severity. In the demo version used by the control group patients, there is no in-app messaging module as well as information such as risk factors, symptoms and intervention recommendations for symptom management.

INTERVENTIONS:
Other: ONKOSIS — ONKOSIS is a mobile phone-based monitoring system in the management of chemotherapy-related symptoms
  Other Names: Mobile Application
  Arms: Intervention Group (ONKOSIS)

SUMMARY:
Mobile health applications open the door to a safe and effective health system. Mobile communication channels and mobile phones not only provide training paths to healthcare professionals, but also provide remote decision support using automated data analysis or the ability to engage in real-time interviews with experts(1). The prevalence of symptoms due to cancer treatment and this adversely affect the quality of life and vital functions of patients and their relatives, and the increase in non-treatment admissions to the hospital. This shows that there is a need for programs where patients can control symptoms related to oncological treatment at home. It is thought that the use of mobile applications can be cost-effective by increasing access to health services and improving diagnosis, treatment and rehabilitation (2). Our single-blind, randomized-controlled, experimental study will be carried out between April 2022 and December 2022 at Kocaeli University Oncology and Palliative Care Center Ambulatory Chemotherapy Unit. The population of the study will consist of chemotherapy patients who applied to the unit and agreed to participate in the study. Based on the calculation made, it was decided to include 212 patients. In this context, it is thought that the mobile-based monitoring system in the management of chemotherapy-related symptoms will contribute to the management of treatment-related symptoms and increase the quality of life in patients receiving chemotherapy.

Expected results from the use of the mobile application;

* reducing the symptom burden,
* improving the quality of life,
* enabling informed changes in clinical practice and care,
* reducing the social and economic burdens of cancer care.

DETAILED DESCRIPTION:
The oncology symptom management system will help patients undergoing cancer treatment manage their symptoms and side effects while going about their daily lives. Therefore, the main customer base consists of patients receiving cancer treatment. However, with the implementation of the application, studies will be carried out in line with the targeted work packages. It is foreseen that the results to be obtained from this will increase the market diversity by integrating the institutions from which cancer treatment patients receive service into the system. For example, improving the quality of life of cancer patients using the application, providing better symptom management in home conditions and reducing the rates of admission to the hospital will reduce the costs of private health insurance companies and increase their profit rates. In addition, if the application is used in the follow-up of patients receiving cancer treatment services from A group private hospitals, it is predicted that institutional satisfaction will increase as well as other added values. It will be possible for private health insurance companies to use the Oncology symptom management system to reduce costs by reducing non-monitoring hospital admissions. In addition, it will be possible for health institutions providing oncology case manager nursing services to use the application in order to increase patient satisfaction and provide patient follow-up. It is planned to provide access to oncology nurses by participating in professional organizations to be held and cooperating with institutions such as the Oncology Nurses Association. It is aimed to use the Oncology Symptom Management System mobile application in our country in symptom management by cancer patients, in patient follow-up by healthcare professionals, and in scientific studies by academics.

ELIGIBILITY:
Inclusion Criteria:

1. Being diagnosed with cancer
2. Receiving first-line cytotoxic chemotherapy

   * Have been scheduled to receive 2, 3, or 4 week chemotherapy protocols (ie, chemotherapy administered in repeated cycles of 14, 21, or 28 days, respectively)
3. To receive at least 3 cycles of chemotherapy
4. To be deemed fit to participate in the research physically/psychologically by the researcher
5. Not having a communication barrier, having the ability to understand and use the mobile application.

Exclusion Criteria:

1. Receiving chemotherapy for the same type of cancer or another type of cancer before being included in the study
2. Patients with treatment protocol changes during chemotherapy will be excluded from participation.
3. Receiving simultaneous radiotherapy during chemotherapy treatment
4. To be programmed to receive a weekly chemotherapy protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2023-06-23 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Changes in quality of life as a result of the intervention | At the end of each cycle of chemotherapy (each cycle can be either 14, 21 or 28 days long) for up to a maximum of 6 cycles of chemotherapy.
  The Nightingale Symptom Rating Scale will be used to evaluate the quality of life of patients using the mobile application compared to the control group. The Nightingale Symptom Rating Scale is a Likert-type quality of life scale used to evaluate the severity of treatment-related symptoms in cancer patients. It includes 38 symptoms frequently reported by cancer patients. The severity of symptoms experienced by patients is measured using five possible numerical responses; where 0 = not at all, 1 = a little, 2 = a little, 3 = quite a lot, and 4 = a lot. High scores indicate that patients' general quality of life or well-being regarding related sub-dimensions is poor.

SECONDARY OUTCOMES:
Evaluation of application to hospital out of monitoring | At the end of chemotherapy, a maximum of 6. cycles (each cycle can be 14, 21 or 28 days)
  Admission to hospital due to chemotherapy side effects during treatment
Assessment of Satisfaction | At the end of chemotherapy, a maximum of 6. cycles (each cycle can be 14, 21 or 28 days)
  App satisfaction score (0-10)
Evaluation of suggested interventions in symptom management | At the end of chemotherapy, up to a maximum of 6. cycles (each cycle can be 14, 21 or 28 days)
  It is aimed to evaluate the effectiveness of the interventions recommended by the patients to manage the symptoms in oncology patients receiving chemotherapy. Efficiency score of the proposed interventions in coping with chemotherapy side effects (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Gülbeyaz Can, Prof, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Ünal ÖNSÜZ, Kocaeli, Kartepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kearney N, McCann L, Norrie J, Taylor L, Gray P, McGee-Lennon M, Sage M, Miller M, Maguire R. Evaluation of a mobile phone-based, advanced symptom management system (ASyMS) in the management of chemotherapy-related toxicity. Support Care Cancer. 2009 Apr;17(4):437-44. doi: 10.1007/s00520-008-0515-0. Epub 2008 Oct 25. PMID 18953579
- [Background] McCann L, Maguire R, Miller M, Kearney N. Patients' perceptions and experiences of using a mobile phone-based advanced symptom management system (ASyMS) to monitor and manage chemotherapy related toxicity. Eur J Cancer Care (Engl). 2009 Mar;18(2):156-64. doi: 10.1111/j.1365-2354.2008.00938.x. PMID 19267731
- [Background] Maguire R, McCann L, Kotronoulas G, Kearney N, Ream E, Armes J, Patiraki E, Furlong E, Fox P, Gaiger A, McCrone P, Berg G, Miaskowski C, Cardone A, Orr D, Flowerday A, Katsaragakis S, Darley A, Lubowitzki S, Harris J, Skene S, Miller M, Moore M, Lewis L, DeSouza N, Donnan PT. Real time remote symptom monitoring during chemotherapy for cancer: European multicentre randomised controlled trial (eSMART). BMJ. 2021 Jul 21;374:n1647. doi: 10.1136/bmj.n1647. PMID 34289996